CLINICAL TRIAL: NCT06928558
Title: Prevalence of Preoperative Anemia in the Oncology Population and Associated Mortality
Brief Title: Preoperative Anemia in the Oncology Population and Associated Mortality
Status: Not yet recruiting | Type: Observational
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Roberto Gonzalez Cornejo, Anesthesiologist, University of Chile
Other Study IDs: Instituto Nacional del Cáncer
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Anemia; Oncologic Surgery
Keywords: Anemia; Oncologic Surgery; Anesthesia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Surgical oncology patients: Oncology patients over 18 years of age, scheduled for surgery with curative intent

SUMMARY:
Anemia is a highly prevalent condition in the surgical population (1, 2). On the other hand, the oncology population is at higher risk of developing anemia due to specific treatments for the disease, such as chemotherapy and radiotherapy. Preoperative anemia has been associated with an increased risk of postoperative morbidity and even mortality (3). Despite this, the prevalence of preoperative anemia in the Chilean oncology population has not been quantified. To answer this question, a retrospective cohort study was designed between January and December 2022 to quantify the prevalence of anemia in the surgical population of the National Cancer Institute. In addition, the impact on morbidity and mortality at 30 days, 6 months, and 1 year will be evaluated. Statistical analysis will be performed using R. Studio Version 2023.09.1+494 (2023.09.1+494).

DETAILED DESCRIPTION:
General Objective:

To quantify the prevalence of preoperative anemia in the National Cancer Institute's oncology surgical population and its impact on postoperative outcomes.

Specific Objectives:

1. To quantify the prevalence of preoperative anemia in the National Cancer Institute's oncology population.
2. To stratify the prevalence of preoperative anemia in the National Cancer Institute's oncology population by severity.
3. To assess 30-day, 6-month, and 1-year mortality in cancer patients with and without anemia in the National Cancer Institute's oncology population.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Oncologic surgery with curative intent

Exclusion Criteria:

* Emergency surgery
* Patients who received a preoperative transfusion
* Patients without a preoperative blood count

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients operated at the National Cancer Institute will be included in a retrospective cohort study between January and December 2022.
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Prevalence of preoperative anemia | 1 year
  To quantify the prevalence of preoperative anemia in the oncology surgical population of the National Cancer Institute and its impact on postoperative outcomes.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sim YE, Abdullah HR. Implications of Anemia in the Elderly Undergoing Surgery. Clin Geriatr Med. 2019 Aug;35(3):391-405. doi: 10.1016/j.cger.2019.04.001. Epub 2019 May 27. PMID 31230739
- [Background] Goodnough LT, Shander A, Spivak JL, Waters JH, Friedman AJ, Carson JL, Keating EM, Maddox T, Spence R. Detection, evaluation, and management of anemia in the elective surgical patient. Anesth Analg. 2005 Dec;101(6):1858-1861. doi: 10.1213/01.ANE.0000184124.29397.EB. PMID 16301274
- [Background] Musallam KM, Tamim HM, Richards T, Spahn DR, Rosendaal FR, Habbal A, Khreiss M, Dahdaleh FS, Khavandi K, Sfeir PM, Soweid A, Hoballah JJ, Taher AT, Jamali FR. Preoperative anaemia and postoperative outcomes in non-cardiac surgery: a retrospective cohort study. Lancet. 2011 Oct 15;378(9800):1396-407. doi: 10.1016/S0140-6736(11)61381-0. Epub 2011 Oct 5. PMID 21982521